CLINICAL TRIAL: NCT01551888
Title: A Phase 2a, Randomized, Open-Label, 2-Way Crossover Study To Determine The Pharmacokinetics, Safety, And Tolerability Of Aclidinium/Formoterol 400/12 µg Fixed Dose Combination Via Almirall Inhaler And Formoterol 12 µg Via Foradil® Aerolizer® In Patients With Moderate To Severe Chronic Obstructive Pulmonary Disease
Brief Title: Pharmacokinetic, Safety and Tolerability Study of Aclidinium/Formoterol Fixed Dose Combination and Formoterol in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LAC-PK-01
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Results first posted 2016-11-23 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclidinium/formoterol 400/12μg FDC (Experimental): Aclidinium/formoterol 400/12μg fixed-dose combination (FDC), one inhalation twice daily (morning and evening) for 4 days, then one inhalation (morning) on Day 5 via the Almirall inhaler
  Interventions: Drug: Aclidinium/formoterol 400/12μg
- Formoterol (Active Comparator): Formoterol 12μg one inhalation twice daily (morning and evening) for 4 days, then one inhalation (morning) on Day 5 via the Foradil® Aerolizer®
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: Aclidinium/formoterol 400/12μg — Aclidinium/formoterol 400/12μg fixed dose combination (FDC), one inhalation twice daily (morning and evening) for 4 days, then one inhalation (morning) on Day 5 via the Almirall inhaler
  Arms: Aclidinium/formoterol 400/12μg FDC
Drug: Formoterol — Formoterol 12 μg one inhalation twice daily (morning and evening) for 4 days, then one inhalation (morning) on Day 5 via the Foradil® Aerolizer®
  Other Names: Foradil® Aerolizer®
  Arms: Formoterol

SUMMARY:
The purpose of this Phase II study is to evaluate the pharmacokinetics, safety, and tolerability of aclidinium/formoterol fixed dose combination (FDC 400/12 μg via the Almirall Inhaler and formoterol 12 μg via the Foradil® Aerolizer®, both administered twice daily for five days to patients with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* Current or former cigarette smokers with a cigarette smoking history of at least 10 pack-years
* A diagnosis of stable moderate to severe COPD and stable airway obstruction as defined by the Global Initiative for Chronic Obstructive Lung Disease guidelines and stable airway obstruction.

Exclusion Criteria:

* Patients who have been hospitalized for an acute COPD exacerbation within three months prior to Screening
* Any respiratory tract infection (including the upper respiratory tract) or COPD exacerbation in the six weeks before Screening
* Patients with any clinically significant respiratory conditions other than COPD
* Clinical history that suggests that the patient has asthma as opposed to COPD
* Chronic use of oxygen therapy ≥ 15 hours/day
* Patients with clinically significant cardiovascular conditions
* Patients with a history of hypersensitivity reaction to inhaled anticholinergics, beta-2 agonists, sympathomimetic amines, or inhaled medications

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (1):
- Forest Investigative Site 001, Spartanburg, South Carolina, United States

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4102&filename=LAC-PK-01_CSRredacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in a single center in the United States
  First patient visit was in January 2012 and last patient visit was in March 2012
Groups:
- Sequence 1: Aclidinium/formoterol 400 μg/12 μg FDC (via the Almirall inhaler) one inhalation twice daily (morning and evening) for 4 days, then one inhalation (morning) for 1 day in Period 1 and, in Period 2, Formoterol 12 μg via the Foradil® Aerolizer®, one inhalation twice daily (morning and evening) for 4 days, then one inhalation (morning) for 1 day
- Sequence 2: Formoterol 12 μg via the Foradil® Aerolizer®, one inhalation twice daily (morning and evening) for 4 days, then one inhalation (morning) for 1 day in Period 1 and, in Period 2, Aclidinium/formoterol 400 μg/12 μg FDC (via the Almirall inhaler) one inhalation twice daily (morning and evening) for 4 days, then one inhalation (morning) for 1 day
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All patients participating in the crossover study
Arm/Group | Overall Study Population
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (7.5)
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Formoterol Plasma Concentration Versus Time Curve (AUC) Over Dosing Interval at Steady State
Description: The standard deviation of the measure is expressed as the coefficient of variation (%)
Time Frame: Day 1: 0, 5, 15 and 30 min and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours (5 min before PM dose) and 5 and 15 min post PM dose; Days 2-4: 0, 5 and 15 min post dose; Day 5: 0, 5, 15 and 30 min and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours (post AM dose)
Population: The pharmacokinetic (PK) analysis population included all patients who completed the study and had evaluable PK parameters
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Groups:
- Formoterol 12 μg: Administered via Foradil® Aerolizer®
- Aclidinium/Formoterol 400/12 μg FDC: Fixed dose combination (FDC) administered via Almirall inhaler
Arm/Group | Formoterol 12 μg | Aclidinium/Formoterol 400/12 μg FDC
Number analyzed (Participants) | 24 | 24
pg*hr/mL | 87.14 (27.8) [0.08 to 2.00] | 85.15 (28.3) [0.08 to 2.00]

2. Primary Outcome: Maximum Formoterol Plasma Drug Concentration (Cmax) at Steady State
Description: The standard deviation of the measure is expressed as the coefficient of variation (%)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Formoterol 12 μg | Aclidinium/Formoterol 400/12 μg FDC
Number analyzed (Participants) | 24 | 24
pg/mL | 14.90 (27.9) [lower limit 27.9] | 16.72 (31.6)

3. Secondary Outcome: Area Under the Formoterol Plasma Concentration Versus Time Curve (AUC) Over Dosing Interval Following a Single Dose
Description: The standard deviation of the measure is expressed as the coefficient of variation (%)
Time Frame: Day 1: 0, 5, 15 and 30 min and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours (5 min before PM dose) and 5 and 15 min post PM dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Formoterol 12 μg | Aclidinium/Formoterol 400/12 μg FDC
Number analyzed (Participants) | 24 | 24
pg*hr/mL | 41.63 (32.2) [0.08 to 2.00] | 42.27 (31.3) [0.08 to 2.00]

4. Primary Outcome: Maximum Formoterol Plasma Drug Concentration (Cmax) Following a Single Dose
Description: The standard deviation of the measure is expressed as the coefficient of variation (%)
Time Frame: Day 1: 0, 5, 15 and 30 min and 1, 1.5, 2, 3, 4, 6, 8, and 12 hours (5 min before PM dose) and 5 and 15 min post PM dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Formoterol 12 μg | Aclidinium/Formoterol 400/12 μg FDC
Number analyzed (Participants) | 24 | 24
pg/mL | 8.23 (39.9) [lower limit 27.9] | 9.55 (39.0)

ADVERSE EVENTS:
Time Frame: Up to study Day 17
Groups:
- Aclidinium/Formoterol 400/12 μg: Fixed dose combination (FDC) administered via Almirall inhaler
Arm/Group | Aclidinium/Formoterol 400/12 μg | Formoterol 12 μg
Serious Adverse Events (participants affected / at risk) | 0/24 | 2/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium/Formoterol 400/12 μg (N=24) | Formoterol 12 μg (N=24)
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the PI will be subject to mutual agreement between the PI and sponsor.